CLINICAL TRIAL: NCT04577781
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of GLPG3970, Administered Orally for 6 Weeks in Adult Subjects With Moderately to Severely Active Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Brief Title: A Study Evaluating the Effects of GLPG3970 Given as an Oral Treatment for 6 Weeks in Adults With Moderately to Severely Active Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Acronym: LADYBUG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG3970-CL-209; 2020-000658-83 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; Rheumatic Diseases; Moderately active rheumatoid arthritis; Severely active rheumatoid arthritis; Joint Diseases; Autoimmune Diseases; Musculoskeletal Diseases; Musculoskeletal and connective tissue disorders
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Rheumatic Diseases; Joint Diseases; Autoimmune Diseases; Musculoskeletal Diseases; Connective Tissue Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG3970 (Experimental): Participants received 400 milligrams (mg) GLPG3970 oral solution, once daily (QD) for a period of 6 weeks.
  Interventions: Drug: GLPG3970
- Placebo (Placebo Comparator): Participants received GLPG3970 matching placebo oral solution, QD for a period of 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG3970 — GLPG3970 powder and solvent for oral solution to be reconstituted prior to use.
  Arms: GLPG3970
Drug: Placebo — Placebo powder and solvent for oral solution to be reconstituted prior to use.
  Arms: Placebo

SUMMARY:
The primary objective of this study was to evaluate the effect of GLPG3970 compared to placebo on the signs and symptoms of Rheumatoid Arthritis (RA) in participants with moderately to severely active RA and an inadequate response to methotrexate (MTX).

ELIGIBILITY:
Key Inclusion Criteria:

1. A body mass index (BMI) between 18-32 kg/m^2, inclusive.
2. Diagnosis of RA ≥6 months prior to screening AND meeting the 2010 American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) criteria of RA AND ACR functional class I-III.
3. Have ≥6 swollen joints (from a swollen joint count evaluated in 66 joints [SJC66]) AND ≥8 tender joints (from a tender joint count evaluated in 68 joints [TJC68]) at screening and at the baseline visit (Visit 1) prior to the first investigational product (IP) dosing.
4. DAS28 (CRP) >3.2 (moderate disease) at screening.
5. Screening serum high sensitivity C-reactive protein (hsCRP) > upper limit of normal (ULN, central laboratory reference: ≤ 5.0 mg/L).
6. Inadequate response to MTX, i.e. treatment-experienced participants who demonstrated inadequate clinical response during treatment with MTX.
7. Have received MTX for ≥6 months and on stable dose (10 to 20 mg/week) of MTX for at least 4 weeks prior to screening and willing to continue on their current stable dose and dosing regimen for the duration of the study.
8. If taking systemic steroids, prednisone equivalent at a dose of ≤10 mg/day and stable for at least 4 weeks prior to the first IP dosing.

Key Exclusion Criteria:

1. Current therapy with any conventional disease-modifying antirheumatic drug (DMARD) other than MTX, including

   1. oral or injectable gold, sulfasalazine, antimalarials, azathioprine, or D-penicillamine within 4 weeks prior to screening,
   2. cyclosporine within 8 weeks prior to screening, and
   3. leflunomide within 3 months prior to screening or a minimum 4 weeks prior to screening if after 11 days of standard cholestyramine therapy.
2. Current or previous treatment with a biologic DMARD (bDMARD). Except for participants who received bDMARDs only in a single clinical study setting:

   1. For whom the last dose of bDMARD ≥6 months prior to screening (12 months for rituximab or other lymphocyte depleting agents), AND;
   2. For whom the bDMARD was effective, without being discontinued due to lack of efficacy.
3. Participants who received an intra-articular or parenteral corticosteroid injection within 4 weeks prior to screening.
4. Participants who received a prior surgical intervention within 12 weeks prior to screening or likely requirement for surgery during the study.
5. Participant has a history of tuberculosis (TB) diagnosis or evidence of active or latent infection with Mycobacterium tuberculosis as defined by one of the following assessments:

   1. Positive QuantiFERON-TB Gold test result at screening, OR
   2. Chest radiograph (posterior anterior view) taken within 12 weeks prior to screening, read by a qualified radiologist or pulmonologist, with evidence of current active TB or old inactive TB.
6. Participant has any active systemic infection within the last 2 weeks prior to first IP dosing, or poorly controlled chronic cardiac, pulmonary or renal disease.
7. Participant has a known or suspected history of or a current immunosuppressive condition, or a history of invasive opportunistic infections (e.g. human immunodeficiency virus [HIV] infection, histoplasmosis, listeriosis, coccidiodmycosis, pneumocystosis, aspergillosis).
8. Participant has a chronic hepatitis B virus (HBV) infection, as defined by persistent HBV surface antigen (HBsAg) positivity. Participant has hepatitis C virus (HCV) infection, as defined by positive HCV antibody at screening and detectable HCV viremia. Participants with positive HCV antibody must undergo reflex HCV ribonucleic acid (RNA) testing, and participants with HCV RNA positivity will be excluded. Participants with positive HCV antibody and negative HCV RNA are eligible.
9. Participant testing positive at screening for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as detected by real time polymerase chain reaction (RT-PCR), participants presenting any signs or symptoms as detected at baseline following careful physical examination (e.g. cough, fever, headaches, fatigue, dyspnea, myalgia, anosmia, dysgeusia, anorexia, sore throat, others) or reporting any signs and symptoms for the 2 preceding weeks, or participants who have been exposed to individuals with confirmed or suspected diagnosis of SARS-CoV-2 within 2 weeks prior to baseline. In addition, any other locally applicable standard diagnostic criteria may also apply to rule out SARS-CoV-2 infection.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Medical Director, Study Director — Galapagos NV
Locations (9):
- Bulgaria (2):
  - Medical Center Teodora, Rousse
  - UMHAT Sv. Ivan Rilski EAD, Sofia
- Georgia (2):
  - Aversi Clinic Ltd, Tbilisi
  - Consilium Medulla-multiprofile clinic Ltd, Tbilisi
- Poland (2):
  - Centrum Medyczne Grunwald, Poznan
  - Centrum Badan Klinicznych S.C., Poznan
- Ukraine (3):
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia
  - Medical Center Clinic of Modern Rheumatology, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted across 4 countries (Georgia, Poland, Bulgaria, and Ukraine). A total of 54 participants were screened, out of which 28 were randomized and treated.
Pre-assignment Details: Participants remained on a stable dose (10 to 20 mg/week) of MTX as background medication.
Period: Overall Study
Arm/Group | GLPG3970 | Placebo
Started | 16 | 12
Completed | 13 | 10
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) consisted of all participants who received at least 1 dose of investigational product.
Groups:
- GLPG3970: Participants received 400 mg GLPG3970 oral solution, QD for a period of 6 weeks.
- Total: Total of all reporting groups
Arm/Group | GLPG3970 | Placebo | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.3) | 41.4 (8.6) | 44.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 12 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 12 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Disease Activity Score Based on 28 Joints C-reactive Protein [DAS28 (CRP)] [Mean (Standard Deviation); unit: Score on a scale] — The DAS28 (CRP) is a derived measurement with differential weighting given to each component such as Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), patient's global assessment of disease activity, and serum CRP level.
  DAS28 (CRP) = 0.56 x square root of TJC28 + 0.28 x square root of SJC28 + 0.36 x Ln[1+CRP(in mg/L)] + 0.014 x patient's disease activity VAS (in mm) + 0.96. A lower score is considered as better disease activity.
  Score on a scale | 6.13 (0.87) | 5.68 (0.88) | 5.93 (0.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DAS-28 (CRP) at Week 6
Description: The DAS28 (CRP) is a derived measurement with differential weighting given to each component such as TJC28, SJC28, patient's global assessment of disease activity, and serum CRP level.
  * TJC28 ranges from 0-28
  * SJC28 ranges from 0-28
  * High sensitivity C-reactive protein (hsCRP) (in mg/L)
  * Patient's disease activity VAS (in mm) (ranges from 0 = best to 100 = worst)
  The DAS28 (CRP) score was calculated using the below formula:
  DAS28 (CRP) = 0.56 x square root of TJC28 + 0.28 x square root of SJC28 + 0.36 x Ln[1+CRP(in mg/L)] + 0.014 x patient's disease activity VAS (in mm) + 0.96. A lower score is considered as better disease activity.
Time Frame: Baseline and Week 6
Population: Full analysis set (FAS) consisted of all randomized participants who had been administered at least 1 dose of investigational product. Participants with available data at specified timepoint were included.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 13 | 10
Score on a scale | -1.29 (0.224) | -1.24 (0.258)
Statistical Analysis 1: Comparison: GLPG3970 vs Placebo; Test type: Superiority; p = 0.885, MMRM — Mixed model repeated measure (MMRM) with treatment-by-visit interaction and baseline-by-visit interaction as fixed effects (with an unstructured variance-covariance matrix); Least Squares (LS) Mean difference = -0.05, 90% CI 2-sided [-0.66 to 0.55], Standard Error of Mean 0.353

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment-Emergent Adverse Events (TEAE) were defined as
  * Any adverse event (AE) with an onset date on or after the IP start date and no later than 14 days after last dose of IP, or worsening of any AE on or after the IP start date.
  * Improvement or no change of any ongoing AEs on or after the IP start date are not considered treatment-emergent. If an AE was ongoing at the time of first IP intake and if there was no change or an improvement in its toxicity grade or its seriousness status, this AE was not considered as treatment-emergent.
  Serious TEAE was defined as a TEAE that
  * Resulted in death and was life-threatening;
  * Required in-patient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly / birth defect;
  * Was medically significant;
Time Frame: From first dose of study drug until end of the study (up to 8 weeks)
Population: Participants in the safety analysis set
Measure: Number; unit: Participants
Groups:
- GLPG3970: Participants received 400 mg GLPG3970 oral solution, QD for a period 6 weeks.
Arm/Group | GLPG3970 | Placebo
Number analyzed (Participants) | 16 | 12
Participants
  TEAE | 6 | 2
  Serious TEAE | 0 | 0
  TEAE leading to death | 0 | 0
  Treatment related TEAE | 4 | 1
  TEAEs leading to study drug discontinuation | 2 | 0

3. Secondary Outcome: Plasma Concentration (Ctrough) of GLPG3970
Description: Ctrough was defined as plasma concentration level at the end of the dosing interval.
Time Frame: Day 15: pre-dose; Day 29: pre-dose; Day 43: pre-dose
Population: Pharmacokinetic analysis set (PKAS) consisted all participants who received at least 1 dose of investigational product with available plasma concentration data. Participants with available plasma concentration at specified time point were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GLPG3970
Number analyzed (Participants) | 11
Nanogram per milliliter
  Day 15: Pre-dose | 95.3 (115)
  Day 29: Pre-dose: number analyzed (Participants) | 9
  Day 29: Pre-dose | 103 (73.8)
  Day 43: Pre-dose: number analyzed (Participants) | 9
  Day 43: Pre-dose | 49.8 (697)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of the study (up to 8 weeks)
Description: Safety analysis set
Arm/Group | GLPG3970 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 6/16 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG3970 (N=16) | Placebo (N=12)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04577781/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04577781/SAP_001.pdf